CLINICAL TRIAL: NCT04912011
Title: The Use of a Mineralocorticoid Receptor Antagonist (Spironolactone) in the Treatment of Pulmonary Fibrosis Associated With SARS-CoV-2 Infection
Brief Title: Mineralocorticoid Receptor Antagonist and Pulmonary Fibrosis in COVID-19.
Acronym: SpiroCOVID19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, Primary Investigator, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0012/100/2020
Record Dates: First submitted 2021-06-01; First posted 2021-06-03 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; spironolactone; pneumonia; fibrosis; SARS-CoV-2; potassium canrenoate
MeSH Terms: conditions — COVID-19; Pneumonia; Fibrosis | interventions — Canrenoic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canrenoate potassium (Experimental): Administration of 200 mg of potassium Canrenoate potassium dissolved in 100 ml of 0.9% sodium chloride intravenously twice a day for 7 days.
  Interventions: Drug: Canrenoate Potassium
- Placebo (Placebo Comparator): Administration of 100 ml of 0.9% sodium chloride intravenously twice a day for 7 days.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Canrenoate Potassium — Intervention: 200 mg of Canrenoate potassium in 100 ml 0,9% NaCl, intravenously twice a day for 7 days.
  Other Names: Investigational Product
  Arms: Canrenoate potassium
Drug: Normal Saline — Placebo: 100 ml 0,9% NaCl, intravenously twice a day for 7 days.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
In December 2019 SARS-CoV-2 virus appeared in the world, mainly appearing as an acute infection of the lower respiratory tract. In March 2020, the World Health Organization (WHO) announced a pandemic in relation to the disease caused by the SARS-CoV-2 virus, known as COronaVIrus Disease 2019 (COVID-19). Since then, the efforts of scientists from around the world have focused on finding the right treatment and vaccine for the new disease. COVID-19 has spread rapidly in a few months, affecting patients in all ages. The disease has a varied course, patients can be 80% asymptomatic, but many develop respiratory failure, complicated by sepsis and ultimately death. One of the possible complications associated with COVID-19 lung involvement is pulmonary fibrosis, leading to chronic breathing difficulties and prolonged disability. No specific mechanisms leading to this phenomenon have been identified in COVID-19, but some information is derived from previous studies on the SARS and MERS epidemic. There have been several reports that the use of spironolactone may be important in preventing pulmonary fibrosis.

The aim of the study is to evaluate the effectiveness of intravenous form of mineralocorticoid receptor antagonist canrenoate potassium (an aldosterone antagonist of the spirolactone group) in the treatment of COVID-19-associated pulmonary fibrosis based on the mechanisms of the immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, 18-90 years of age.
2. Patient requiring oxygen therapy, SpO2 <94%.
3. Confirmed COVID-19 infection.
4. At least one risk factor for increased mortality in the course of COVID-19: currently published in the literature e.g. smoking, hypertension, diabetes, cardiovascular disease.
5. Documented informed consent according to ICH-GCP and national regulations.

Exclusion Criteria:

1. Chronic bronchitis, emphysema, interstitial lung disease, or other history of lung disease.
2. Contraindications to the use of spironolactone.
3. Hypersensitivity to spironolactone or any of the excipients.
4. Pregnant patients (pregnancy test will be performed in every patient of reproductive age) and during lactation.
5. Patients with mental illness or dementia who are unable to give informed consent to the examination.
6. ARDS caused by another viral infection (SARS-CoV-2 negative).
7. ARDS from other causes/trauma.
8. Ionic disorders: hyperkalemia, hyponatraemia.
9. Adrenal crisis.
10. Acute and chronic renal failure, creatinine clearance less than 30 ml/min.
11. Anuria.
12. Porphyria.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation | 30 days
  Duration of invasive mechanical ventilation via endotracheal intubation or tracheotomy
Passive oxygen therapy | 30 days
  Duration of passive oxygen therapy

SECONDARY OUTCOMES:
ICU LOS | 30 days
  Intensive Care Unit length of stay (LOS).
Hospital LOS | 90 days
  Total hospital length of stay (LOS).
Chest CT | 90 days
  Assessment of the dynamics of recovery of changes in chest CT at 3 months.
Lung ultrasound_7 | 7 days
  Assessment of the dynamics of recovery of changes in lung ultrasound at 7 days.
Lung ultrasound_30 | 30 days
  Assessment of the dynamics of recovery of changes in lung ultrasound at 30 days.
Mortality_30 | 30 days
  Assessment of mortality at 30 days.
Mortality_90 | 90 days
  Assessment of mortality at 90 days.
IL-1β level change. | 7 days
  Evaluation of the degree of change of the level of pro-inflammatory cytokine IL-1β.
IL-2 level change. | 7 days
  Evaluation of the degree of change of the level of pro-inflammatory cytokine IL-2.
IL-6 level change. | 7 days
  Evaluation of the degree of change of the level of pro-inflammatory cytokine IL-6.
IL-33 level change. | 7 days
  Evaluation of the degree of change of the level of pro-inflammatory cytokine IL-33.
TNFα level change. | 7 days
  Evaluation of the degree of change of the level of pro-inflammatory cytokine TNFα.
6MWT | 30 days
  Six minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna L Kotfis, MD, PhD, Principal Investigator — Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechowicz K, Drozdzal S, Machaj F, Rosik J, Szostak B, Zegan-Baranska M, Biernawska J, Dabrowski W, Rotter I, Kotfis K. COVID-19: The Potential Treatment of Pulmonary Fibrosis Associated with SARS-CoV-2 Infection. J Clin Med. 2020 Jun 19;9(6):1917. doi: 10.3390/jcm9061917. PMID 32575380
- [Background] Kotfis K, Lechowicz K, Drozdzal S, Niedzwiedzka-Rystwej P, Wojdacz TK, Grywalska E, Biernawska J, Wisniewska M, Parczewski M. COVID-19-The Potential Beneficial Therapeutic Effects of Spironolactone during SARS-CoV-2 Infection. Pharmaceuticals (Basel). 2021 Jan 17;14(1):71. doi: 10.3390/ph14010071. PMID 33477294